CLINICAL TRIAL: NCT02151006
Title: Does DHEA Improve Pregnancy Rate in Women Undergoing IVF/ICSI With Expected Poor Ovarian Response According to the Bologna Criteria? A Randomized Controlled Study
Brief Title: Does Dehydro Epiandrosterone (DHEA) Improve Pregnancy Rate in Women Undergoing IVF/ICSI With Expected Poor Ovarian Response?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sub 2
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Subfertility
Keywords: DHEA; IVF; ICSI
MeSH Terms: conditions — Infertility | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHEA (Active Comparator): women will receive DHEA 6 weeks before starting IVF/ICSI
  Interventions: Drug: DHEA
- Control (No Intervention)

INTERVENTIONS:
Drug: DHEA
  Arms: DHEA

SUMMARY:
140 women with expected poor ovarian response undergoing IVF/ICSI will be randomly divided into 2 groups using computer generated random numbers . Group 1 ( study group) will receive DHEA 25 mg ( DHEA 25mg, Natrol , USA) t.d.s daily for 12 weeks before starting IVF/ICSI cycle. Group 2 ( control group) will not receive DHEA. Patients included in the study will be subjected to full history taking and clinical examination. On the second day of menstruation serum FSH, LH, Prolactin and Oestradiol will be assessed and the antral follicular count (AFC) will be assessed using a vaginal ultrasound scan. AFC will be defined as the number of follicles measuring 3-10mm.

All patients will have gonadotropin antagonist protocol with Human menopausal gonadotrophin (HMG) stimulation until the day of (Human chorionic gonadotrophin (HCG) administration. On the day of HCG administration, ovarian ultrasound scan will be performed using a transvaginal probe. Oocytes will be aspirated 34-36 hours after HCG administration. Oocytes will be fertilized and embryos will be transferred. Both groups will be compared regarding the proportion of pregnancy.

DETAILED DESCRIPTION:
The study will be conducted in Cairo university hospitals and Dar Al-Teb Infertility and Assisted conception center, Giza Egypt. All patients attending the centre will be evaluated for their expected ovarian response.Patients fulfilling the Bologna criteria definition of poor ovarian response will be invited to participate in the study and to sign informed consent forms. The invitation will include a clear full explanation of the study.

140 women will be randomly divided into 2 groups using computer generated random numbers. Group 1 ( study group) will include 70 women who will receive DHEA 25 mg t.d.s ( DHEA®, Natrol , USA) twice daily for 12 weeks before starting IVF/ICSI cycle. Group 2 will include 70 women who will not receive DHEA and will serve as the control group. All women fulfilling the inclusion criteria will be invited to participate in the study. A written informed consent will be taken and only women signing the consent will be included in the study.

Patients included in the study will be subjected to full history taking and clinical examination including general, abdominal and gynecological examination. This will be followed by a vaginal ultrasound scan to assess uterus, ovaries and any pelvic masses.

On the second day of menstruation serum FSH, LH, Prolactin and Oestradiol will be assessed and the antral follicular count (AFC) will be assessed using a vaginal ultrasound scan. AFC will be defined as the number of follicles measuring 3-10mm.

The stimulation protocol will start on day 2 using 450-300 IU HMG ( Merional® IBSA, Lugano, Switzerland) and GnRH antagonist, cetrorelix (Cetrotide® Merck Serono, Darmstadt, Germany) 0.025 mg daily. Gonadotropins will be administered for 4 to 5 days, after which the dose will be adjusted according to the ovarian response. The ovarian response will be monitored by transvaginal ultrasound and serum E2 levels. When three or more follicles reached a maximum diameter of 16 mm, highly purified HCG 5000 or 10,000 IU (Choriomon ®IBSA) will be administered. The procedure will be cancelled if less than 3 follicles 16 mm in size are present 12 days after starting gonadotropins despite doses reaching 450 IU. The cycle will be also cancelled if there is risk of ovarian hyperstimulation like massive ovarian enlargement or serum estradiol exceeds 3000pg/L Transvaginal oocyte retrieval will be performed 34-36 h after the administration of HCG. Oocytes will be fertilized either via IVF or ICSI based on the couple's history. Fertilization will be assessed 16-18 h after IVF or ICSI . Embryos will be transferred on Day 3 or 5. Vaginal tablets containing progesterone (Prontogest® IBSA) 400 mg/day will be given when fertilization is confirmed. A pregnancy test will be done 2 weeks after embryo transfer. For patients with a positive pregnancy test, progesterone is to be continued for an additional 4 weeks. Clinical pregnancy will be defined as Visualization of an intrauterine gestational sac 5 weeks after embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing IVF/ICSI treatment with expected poor ovarian response according to the Bologna criteria

Exclusion Criteria:

* Women with BMI >35 Kg/M2
* Women with a single ovary
* Known allergy to DHEA
* Diabetic women on insulin as insulin lowers DHEA levels and might reduce the effectiveness of DHEA supplements

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy | 5 weeks after embryo transfer
  Sonographic detection of a gestational sac

SECONDARY OUTCOMES:
Number of oocytes retrieved | one hour after ovum pick up
Number of formed embryos | 3 days after ovum pick up
Quality of formed embryos | 3 days after ovum pick up

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed MM Kotb, MD, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Cairo University Hospitals, Cairo
  - Dar AlTeb subfertility centre, Giza

REFERENCES:
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041
- [Background] Barad D, Brill H, Gleicher N. Update on the use of dehydroepiandrosterone supplementation among women with diminished ovarian function. J Assist Reprod Genet. 2007 Dec;24(12):629-34. doi: 10.1007/s10815-007-9178-x. Epub 2007 Dec 11. PMID 18071895
- [Background] Casson PR, Lindsay MS, Pisarska MD, Carson SA, Buster JE. Dehydroepiandrosterone supplementation augments ovarian stimulation in poor responders: a case series. Hum Reprod. 2000 Oct;15(10):2129-32. doi: 10.1093/humrep/15.10.2129. PMID 11006185
- [Background] Gleicher N, Weghofer A, Barad DH. The role of androgens in follicle maturation and ovulation induction: friend or foe of infertility treatment? Reprod Biol Endocrinol. 2011 Aug 17;9:116. doi: 10.1186/1477-7827-9-116. PMID 21849061
- [Derived] Kotb MM, Hassan AM, AwadAllah AM. Does dehydroepiandrosterone improve pregnancy rate in women undergoing IVF/ICSI with expected poor ovarian response according to the Bologna criteria? A randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2016 May;200:11-5. doi: 10.1016/j.ejogrb.2016.02.009. Epub 2016 Feb 21. PMID 26963897